CLINICAL TRIAL: NCT07034547
Title: Effect of Botulinum Toxin Type A on Functionality and Quality of Life in Children and Adolescents With Spastic Hemiparetic Cerebral Palsy GMFCS I-II at Teletón Santiago: A Prospective Single-Group Trial
Brief Title: Effect of Botulinum Toxin Type A on Motor Function in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Teletón Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TeletonChile
Record Dates: First submitted 2025-05-27; First posted 2025-06-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Palsy (CP); Spasticity Due to Cerebral Palsy; Hemiparesis
Keywords: botulinum toxin; quality of life; Physical Functional Performances
MeSH Terms: conditions — Cerebral Palsy; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Children Aged 8-17 With Spastic Hemiparetic Cerebral Palsy Treated With Botulinum Toxin Type A
  Interventions: Procedure: Botulinum toxin infiltration

INTERVENTIONS:
Procedure: Botulinum toxin infiltration — Botulinum toxin is a medication that is injected directly into the muscles selected by a physiatrist, based on a clinical evaluation. The doses are determined according to the clinical condition of the spasticity, the patient's age, and weight. The procedure is performed under deep sedation and uses ultrasound and electrostimulation to ensure greater safety and precision.

SUMMARY:
Project Identification and Researchers Title: "Changes in functionality and quality of life when applying the botulinum toxin type A infiltration protocol in children and adolescents with cerebral palsy of the spastic hemiparesis type GMFCS I and II, from the Teletón Institute Santiago: A prospective single-group trial."

This project is led by a group of physiatrists from the Teletón Institute, along with a team of co-investigators specialized in kinesiology, occupational therapy, and nursing.

Study Relevance The study aims to generate scientific evidence on the effectiveness of the BoNT-A infiltration protocol in the functionality and quality of life of children with spastic hemiparesis. The results could optimize therapeutic interventions at the Teletón Institute, improve patient well-being, and expand the coverage of therapeutic services for spasticity.

Problem Statement Cerebral palsy (CP) is the most common motor disability in childhood, with an estimated prevalence of 1.6 per 1,000 live births in developed countries and between 1 and 2 per 1,000 live births in Chile. Spastic CP requires multidisciplinary management, including BoNT-A infiltration. Although BoNT-A has been shown to reduce spasticity, there is a gap in knowledge regarding its impact on overall functionality and quality of life.

Research Question What changes occur in functionality and quality of life when applying the BoNT-A infiltration protocol from the Teletón Institute Santiago in children aged 8 to 17 years, diagnosed with cerebral palsy of the spastic hemiparesis type GMFCS I and II?

Study Objectives General Objective: To compare the results in functionality and quality of life before BoNT-A infiltration, at 4 weeks, and at 12 weeks, in children and adolescents diagnosed with cerebral palsy of the spastic hemiparesis type GMFCS I and II.

Specific Objectives: To evaluate the effect of the infiltration protocol on the functionality of the upper and lower limbs, and on the quality of life of the children and their families.

Hypothesis The BoNT-A infiltration protocol has a positive effect on the functionality of the upper and lower limbs and on the quality of life of children with spastic cerebral palsy.

Method The study is a prospective single-group trial, following participants over time to compare the results of the BoNT-A infiltration protocol. The target population includes children with spastic hemiparesis cerebral palsy GMFCS I-II referred to the botulinum toxin infiltration clinic at the Teletón Institute Santiago. A non-probabilistic convenience sampling will be used, selecting individuals who meet the inclusion and exclusion criteria.

Procedure Patients will be selected and evaluated before infiltration, at 4 weeks, and at 12 weeks post-infiltration. The infiltration will be performed under ultrasound and electrostimulation guidance. Evaluations will include functionality and quality of life scales, such as the Ashworth Scale, Tardieu Scale, Bilan 400 Points Functional Hand Scale, GMFM-88, KIDSCREEN-27, and Goal Attainment Scale.

Data Collection Data collection will be carried out through clinical record review, clinical observation, and application of scales. A homologation protocol will be implemented among operators to standardize the use of the scales.

Variables Variables include age, sex, laterality, GMFCS, infiltrated muscles, infiltration dose, educational level, participation in a school integration program, physical activity, manual functionality, lower limb functionality, quality of life, and goal attainment.

Statistical Analysis A database will be created in Microsoft Excel, and qualitative and quantitative variables will be analyzed. Chi-square tests, repeated measures ANOVA, and Friedman tests will be used to compare measurements over time.

Ethical Considerations The study complies with ethical principles of scientific validity, social utility, researcher competence, favorable risk-benefit ratio, equitable selection of subjects, informed consent, and protection of the privacy and confidentiality of participants.

ELIGIBILITY:
Inclusion Criteria:

* Spastic hemiparesis type Cerebral Palsy
* Gross Motor Classification System I-II
* Age 8 to 17 years (based on validation ages for scales to be used)
* Minimum of 6 months since last botulinum toxin injection
* Informed consent signed by legal guardian and assent from users aged 12 to 17 years

Exclusion Criteria:

* Cognitive impairment that prevents following instructions for functional assessments
* Limitation of joint range not caused by spasticity
* Patients diagnosed with other diseases causing spasticity, different from cerebral palsy
* Patients with other neuromuscular diseases

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Bilan 400 Points Functional Hand Scale | Baseline, 4 weeks, and 12 weeks after intervention
  The Bilan 400 Points Functional Hand Scale is an assessment tool used to measure hand functionality in patients with neuro-musculoskeletal disabilities. This scale is primarily applied to children and adolescents aged 7 to 17 years and evaluates four key dimensions: hand mobility, grip strength, monomanual grasp and object displacement, and bimanual function. Each of these dimensions is scored out of 100 points, totaling 400 points. The scale is useful for quantifying the degree of use of an injured hand and for objectifying the impact of therapeutic interventions. In the Bilan 400 Points Functional Hand Scale, higher scores (close to 400) indicate good or normal hand functionality, while lower scores (close to 0) reflect very limited or severely impaired functionality.
Gross Motor Function Measure (GMFM-88). D and E dimensions | Baseline, 4 weeks, and 12 weeks after intervention
  The GMFM-88 is a standardized tool for assessing changes in gross motor function in children with cerebral palsy. It includes 88 items across five dimensions. Dimensions D and E focus on standing and walking-related tasks. Dimension D evaluates the ability to stand independently, including standing on one leg and transitioning from sitting to standing. Dimension E assesses walking, running, and jumping, such as walking forward, running, and jumping over obstacles. Each item is scored from 0 to 3. Higher scores (close to 100%) indicate better gross motor function and greater independence, while lower scores (close to 0%) reflect significant limitations in performing the evaluated tasks.
KIDSCREEN-27 | Baseline and 12 weeks after intervention
  The KIDSCREEN-27 is a mid-length questionnaire designed to assess health-related quality of life (HRQoL) in children and adolescents aged 8-18. It includes 27 items across five dimensions: physical well-being, psychological well-being, autonomy and parent relations, social support and peer relations, and school environment. It is ideal when HRQoL is relevant but not the main focus of a study, or when the full version is too long. Each item uses a 5-point Likert scale to measure frequency or intensity of experiences. Responses are converted to scores from 0 (poorest HRQoL) to 100 (best HRQoL). Higher scores indicate better perceived quality of life in each dimension.
Goal Attainment Scale | Baseline and 12 weeks after intervention
  The Goal Attainment Scale (GAS) is an individualized assessment tool used to document and score the extent to which a patient achieves their personal goals during an intervention. Each patient sets unique goals, which are formulated using the SMART approach (specific, measurable, achievable, relevant, and time-bound). These goals are rated on a five-point scale: +2 indicates the outcome was much better than expected, +1 somewhat better, 0 exactly as expected, -1 somewhat less than expected, and -2 much worse than expected. This standardized scoring allows for statistical analysis of results and helps tailor interventions to the individual needs of the patient. An average score close to 0 indicates that goals were achieved as planned, while positive values reflect better-than-expected performance and negative values indicate underperformance.

SECONDARY OUTCOMES:
Goniometry | Baseline, 4 weeks, and 12 weeks after intervention
  Goniometry is a technique used to measure the range of motion of joints. It is based on measuring joint mobility angles, and its results help identify joint limitations. Ranges of motion are classified as active, passive, or assisted, depending on the degree of patient involvement in the movement. The values obtained are expressed in degrees (°), and each joint has a normal reference range. For example, elbow flexion typically ranges from 0° to 150°. Values within the normal range indicate adequate functional mobility; values below may reflect stiffness, contractures, or limitations, while values above the expected range may suggest hypermobility or joint instability.
Ashworth Scale | Baseline, 4 weeks, and 12 weeks after intervention
  The Ashworth Scale is a diagnostic tool used to measure muscle tone in patients with spasticity. It assigns a score from 0 to 4 based on the resistance to passive movement of a joint. The scores are: 0: No increase in muscle tone, 1: Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion, 2: More marked increase in muscle tone through most of the range of motion, but the affected part is easily moved, 3: Considerable increase in muscle tone, passive movement difficult, 4: Affected part rigid in flexion or extension.
Tardieu Scale | Baseline, 4 weeks, and 12 weeks after intervention
  The Tardieu Scale is used to assess spasticity in patients with neurological conditions by evaluating muscle response at different stretch speeds and measuring the spasticity angle. It includes two components: the quality of muscle reaction and the angle of reaction. The quality is scored from 0 to 5, where 0 means no resistance, 1 slight resistance, 2 a clear stop with release, 3 a sustained or clonic contraction under 10 seconds, 4 sustained over 10 seconds, and 5 a fixed joint. The angle of reaction (R1) is the point of first resistance during a fast stretch and is compared to the maximum passive range (R2). A greater difference between R2 and R1 indicates more dynamic spasticity, while similar values suggest a fixed contracture.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Teleton Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared, as the participants belong to a vulnerable population and the information is considered sensitive and not appropriate for public dissemination